CLINICAL TRIAL: NCT05685225
Title: Safety and Efficacy of Naltrexone/Acetaminophen for the Acute Treatment of Migraine: A Single-Site, Phase 2 Randomized Trial
Brief Title: Single-Site Study of Naltrexone/Acetaminophen for the Acute Treatment of Migraine: A Phase 2 Randomized Trial
Acronym: AT-06
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No participants enrolled; study suspended due to recruitment challenges.
Sponsor: Allodynic Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AT-06
Record Dates: First submitted 2022-12-27; First posted 2023-01-17 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Migraine
Keywords: Naltrexone; Acetaminophen; Acute migraine; Low-dose naltrexone; Anxiety
MeSH Terms: conditions — Migraine Disorders; Anxiety Disorders | interventions — Acetaminophen

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind, Placebo-Controlled, Parallel-Group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Stage 1: Naltrexone/Acetaminophen (Experimental): One dose for a Qualifying Migraine Attack
  Interventions: Drug: Stage 1: Naltrexone/Acetaminophen
- Stage 1: Naltrexone (Active Comparator): One dose for a Qualifying Migraine Attack
  Interventions: Drug: Stage 1: Naltrexone
- Satge 1: Acetaminophen (Active Comparator): One dose for a Qualifying Migraine Attack
  Interventions: Drug: Stage 1: Acetaminophen
- Stage 1: Placebo (Placebo Comparator): One dose for a Qualifying Migraine Attack
  Interventions: Drug: Stage1: Placebo
- Stage 2: Naltrexone/Acetaminophen-high dose (Experimental): One dose for a qualifying migraine attack
  Interventions: Drug: Stage 2: Naltrxone/Acetaminophen high dose
- Stage 2: Naltrexone/Acetaminophen-medium dose (Experimental): One dose for a qualifying migraine attack
  Interventions: Drug: Stage 2: Naltrexone/Acetaminophen medium dose
- Stage 2: Naltrexone/Acetaminophen-low dose (Experimental): One dose for a qualifying migraine attack
  Interventions: Drug: Stage 2: Naltrxone/Acetaminophen low dose
- Stage 2: Placebo (Placebo Comparator): One dose for a qualifying migraine attack
  Interventions: Drug: Stage 2: Placebo

INTERVENTIONS:
Drug: Stage 1: Naltrexone/Acetaminophen — Combination
  Other Names: ALLOD-2
  Arms: Stage 1: Naltrexone/Acetaminophen
Drug: Stage 1: Naltrexone — Naltrexone alone
  Arms: Stage 1: Naltrexone
Drug: Stage 1: Acetaminophen — Acetaminophen alone
  Arms: Satge 1: Acetaminophen
Drug: Stage1: Placebo — Matching placebo
  Arms: Stage 1: Placebo
Drug: Stage 2: Naltrxone/Acetaminophen high dose — Combination high dose
  Other Names: ALLOD-2
  Arms: Stage 2: Naltrexone/Acetaminophen-high dose
Drug: Stage 2: Naltrexone/Acetaminophen medium dose — Combination medium dose
  Other Names: ALLOD-2
  Arms: Stage 2: Naltrexone/Acetaminophen-medium dose
Drug: Stage 2: Naltrxone/Acetaminophen low dose — Combination low dose
  Other Names: ALLOD-2
  Arms: Stage 2: Naltrexone/Acetaminophen-low dose
Drug: Stage 2: Placebo — Matching Placebo
  Arms: Stage 2: Placebo

SUMMARY:
* This two-stage clinical trial will assess a novel combination therapy for acute migraine. In Stage 1 (factorial), participants will receive the combination, each individual component, or placebo. In Stage 2 (dose-finding), they will test three doses of the combination. Before both stages, participants will complete a run-in period, documenting a migraine attack without study medication. They will then treat one migraine attack in each stage.
* 4 visits
* Requirements: Migraine Diagnosis. BMI below 34. Read, write, and speak English. No opioids, marijuana, benzodiazepines, or excessive alcohol.

DETAILED DESCRIPTION:
This study evaluating naltrexone-acetaminophen in the acute treatment of migraine.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18 to 75 years, inclusive.
2. At least 1-year of history of migraine with or without aura as defined by the International Classification of Headache Disorders 3rd edition 17 (ICHD-3).
3. Migraine onset before age 50 years.
4. Read, write, and speak English
5. BMI Higher than 20 and Lower than 34
6. The female subject who is premenopausal or postmenopausal less than one year or have not had surgical sterilization (i.e., tubal ligation, partial or complete hysterectomy) must have a negative urine pregnancy test, be non-lactating, and commit to using two methods of adequate and reliable contraception throughout the study and for 28 days after taking the last dose of the study medication (e.g., barrier with an additional spermicidal, intra- uterine device, hormonal contraception). Male subjects must be surgically sterile (the procedure occurred greater than 6 months before the Screening Visit) or commit to using two different birth control methods during the study and for 28 days after the last dose of the study medication.

Exclusion Criteria:

1. Pregnant or nursing women or those planning a pregnancy.
2. Used opioids (including methadone and buprenorphine), barbiturate-containing medications, muscle relaxants, or benzodiazepines within 3 months prior to screening.
3. Used any recreational drugs in the past 3 months.
4. Use of medications to treat headaches more than 10 days per month in the past 3 months or use of any pain medication for other pain syndromes for more than 10 days per month.
5. Uncontrolled cardiovascular or cerebrovascular disease or a history of heart failure, atrial fibrillation, or myocardial infarction.
6. Uncontrolled hypertension (systolic/diastolic blood pressure ˃ 140/90 mmHg) or diabetes.
7. Immediate family members or same household members participating in the study.
8. Site personnel, their friends, and family.
9. Abnormal laboratory or ECG results.

   1. Aspartate transaminase (AST/SGOT), alanine transaminase (ALT/SGPT), or alkaline Phosphatase ≥ 1.5 x Upper Limit of Normal (ULN). creatinine ≥ 1.5 x ULN.
   2. BBB or intraventricular conduction defect with a QRS duration ≥ 150 msec. ST-T wave abnormalities.
   3. Hemoglobin < 10 g/dL
   4. Neutrophil count ≤ 1000/μL
   5. Cholesterol ≥ 300 mg/dL
   6. Triglycerides ≥ 500 mg/dL Additional exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-01-31 (Actual); Primary Completion 2025-12-02 (Actual); Study Completion 2025-12-02 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with acute migraine who achieved freedom from pain after dosing | 2 hours after dosing
  Freedom from pain is defined as the absence of headache pain from moderate or severe pain at baseline, without the use of rescue medication. The pain is measured on a 4-point scale, with 0 indicating no pain, 1 for mild pain, 2 for moderate pain, and 3 for severe pain.
Proportion of subjects with acute migraine who achieved freedom from migraine's Most Bothersome Symptoms (MBS) after dosing | 2 hours after dosing
  MBS freedom is defined as the absence of the identified Most Bothersome Symptom (MBS), which can be nausea, photophobia, or phonophobia. The MBS is measured on a binary scale, either absent or present.

SECONDARY OUTCOMES:
Proportion of subjects with acute migraine who achieved pain relief | 2 hours after dosing
  Pain relief is defined as a reduction in headache pain severity from moderate or severe to mild or no headache pain.
Proportion of subjects with acute migraine who achieved freedom from photophobia | 2 hours after dosing
  Freedom from photophobia is defined as absence of photophobia
Proportion of subjects with acute migraine who achieved freedom from phonophobia | 2 hours after dosing
  Freedom from phonophobia is defined as absence of phonophobia
Proportion of subjects with acute migraine who achieved freedom from nausea | 2 hours after dosing
  Freedom from nausea is defined as absence of nausea
Proportion of subjects with acute migraine who achieved sustained pain relief from 2 to 24 hours | 2 to 24 hours
  Sustained pain relief is defined as the reduction of headache pain severity from moderate or severe intensity to mild without the use of rescue medication.
The proportion of subjects with acute migraine who achieved sustained pain freedom from 2 to 24 hours | 2 to 24 hours
  Sustained pain freedom is defined as the absence of any headache pain of any intensity without the use of rescue medication.
Functional disability at 2 hours | 2 hours after dosing
  Functional disability refers to the inability to perform activities of daily living or work tasks to a normal level due to physical, mental, or sensory impairments. It is measured on a scale of 0 to 3, where 0 indicates normal function and 3 indicates the need for bedrest due to severe impairment.
Functional disability at 24 hours | 24 hours after dosing
  Functional disability refers to the inability to perform activities of daily living or work tasks to a normal level due to physical, mental, or sensory impairments. It is measured on a scale of 0 to 3, where 0 indicates normal function and 3 indicates the need for bedrest due to severe impairment.
Use of rescue medications within 24 hours | within 24 hours
  Rescue medication use refers to the use of an additional medication to treat the current migraine.
Pain relapse within 48 hours | within 48 hours
  Pain relapse refers to the reappearance of headache pain of any severity when the subject had been free of pain 2 hours after dosing.

OTHER OUTCOMES:
Hamilton Anxiety Rating Scale score | Baseline (Randomization Visit) to 2 hours after dosing
  The Hamilton Anxiety Rating Scale is a validated assessment tool for measuring anxiety symptoms. The scale consists of fourteen items designed to assess the severity of anxiety on a scale of zero to four, with four being the most severe.
Hamilton Anxiety Rating Scale score | Baseline (Randomization Visit) to 24 hours after dosing
  The Hamilton Anxiety Rating Scale is a validated assessment tool for measuring anxiety symptoms. The scale consists of fourteen items designed to assess the severity of anxiety on a scale of zero to four, with four being the most severe.
Self-reported overall sense of wellbeing | 2 hours after dosing
  Self-reported overall sense of wellbeing (physical and emotional) is a subjective measurement that reflects an individual's perception of their physical and emotional health. It is typically assessed on a 4-point scale, ranging from 0 (Poor) to 3 (Superb), with 1 (Okay) and 2 (Good) representing intermediate levels of wellbeing. This measurement considers factors such as physical pain, positive emotions, life satisfaction, stress management, and the absence of negative emotions like depression and anxiety.
Self-reported hurt feelings score | 2 hours after dosing
  Self-reported hurt feelings on a 4-point scale: (0=Not at all, 1=Slightly, 2=Moderate, 3=Extremely).
Self-reported tense feelings score | 2 hours after dosing
  Self-reported tense feelings on a 4-point scale: (0=Not at all, 1=Slightly, 2=Moderate, 3=Extremely).

CONTACTS AND LOCATIONS:
Overall Officials: Annette C Toledano, MD, Study Director — Allodynic Therapeutics, Inc; Natalia Belikova, MD PhD, Principal Investigator — Keystone Clinical Research
Locations (1):
- Keystone Clinical Research, North Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lipton RB, Baggish JS, Stewart WF, Codispoti JR, Fu M. Efficacy and safety of acetaminophen in the treatment of migraine: results of a randomized, double-blind, placebo-controlled, population-based study. Arch Intern Med. 2000 Dec 11-25;160(22):3486-92. doi: 10.1001/archinte.160.22.3486. PMID 11112243
- [Background] Wieseler J, Ellis A, McFadden A, Stone K, Brown K, Cady S, Bastos LF, Sprunger D, Rezvani N, Johnson K, Rice KC, Maier SF, Watkins LR. Supradural inflammatory soup in awake and freely moving rats induces facial allodynia that is blocked by putative immune modulators. Brain Res. 2017 Jun 1;1664:87-94. doi: 10.1016/j.brainres.2017.03.011. Epub 2017 Mar 16. PMID 28322750
- [Background] Marmura MJ, Silberstein SD, Schwedt TJ. The acute treatment of migraine in adults: the american headache society evidence assessment of migraine pharmacotherapies. Headache. 2015 Jan;55(1):3-20. doi: 10.1111/head.12499. PMID 25600718
- [Background] Hutchinson MR, Zhang Y, Brown K, Coats BD, Shridhar M, Sholar PW, Patel SJ, Crysdale NY, Harrison JA, Maier SF, Rice KC, Watkins LR. Non-stereoselective reversal of neuropathic pain by naloxone and naltrexone: involvement of toll-like receptor 4 (TLR4). Eur J Neurosci. 2008 Jul;28(1):20-9. doi: 10.1111/j.1460-9568.2008.06321.x. PMID 18662331
- [Background] Nicotra L, Loram LC, Watkins LR, Hutchinson MR. Toll-like receptors in chronic pain. Exp Neurol. 2012 Apr;234(2):316-29. doi: 10.1016/j.expneurol.2011.09.038. Epub 2011 Oct 6. PMID 22001158
- [Background] Ellis A, Wieseler J, Favret J, Johnson KW, Rice KC, Maier SF, Falci S, Watkins LR. Systemic administration of propentofylline, ibudilast, and (+)-naltrexone each reverses mechanical allodynia in a novel rat model of central neuropathic pain. J Pain. 2014 Apr;15(4):407-21. doi: 10.1016/j.jpain.2013.12.007. Epub 2014 Jan 9. PMID 24412802
- [Background] Lewis SS, Loram LC, Hutchinson MR, Li CM, Zhang Y, Maier SF, Huang Y, Rice KC, Watkins LR. (+)-naloxone, an opioid-inactive toll-like receptor 4 signaling inhibitor, reverses multiple models of chronic neuropathic pain in rats. J Pain. 2012 May;13(5):498-506. doi: 10.1016/j.jpain.2012.02.005. Epub 2012 Apr 20. PMID 22520687
- [Background] Wang X, Zhang Y, Peng Y, Hutchinson MR, Rice KC, Yin H, Watkins LR. Pharmacological characterization of the opioid inactive isomers (+)-naltrexone and (+)-naloxone as antagonists of toll-like receptor 4. Br J Pharmacol. 2016 Mar;173(5):856-69. doi: 10.1111/bph.13394. Epub 2016 Feb 4. PMID 26603732
- [Background] Selfridge BR, Wang X, Zhang Y, Yin H, Grace PM, Watkins LR, Jacobson AE, Rice KC. Structure-Activity Relationships of (+)-Naltrexone-Inspired Toll-like Receptor 4 (TLR4) Antagonists. J Med Chem. 2015 Jun 25;58(12):5038-52. doi: 10.1021/acs.jmedchem.5b00426. Epub 2015 Jun 5. PMID 26010811
- [Background] Roberts ID, Krajbich I, Way BM. Acetaminophen influences social and economic trust. Sci Rep. 2019 Mar 11;9(1):4060. doi: 10.1038/s41598-019-40093-9. PMID 30858394
- [Background] Dewall CN, Macdonald G, Webster GD, Masten CL, Baumeister RF, Powell C, Combs D, Schurtz DR, Stillman TF, Tice DM, Eisenberger NI. Acetaminophen reduces social pain: behavioral and neural evidence. Psychol Sci. 2010 Jul;21(7):931-7. doi: 10.1177/0956797610374741. Epub 2010 Jun 14. PMID 20548058
- [Background] Wardle MC, Bershad AK, de Wit H. Naltrexone alters the processing of social and emotional stimuli in healthy adults. Soc Neurosci. 2016 Dec;11(6):579-91. doi: 10.1080/17470919.2015.1136355. Epub 2016 Jan 22. PMID 26710657
- [Background] Devlen J. Anxiety and depression in migraine. J R Soc Med. 1994 Jun;87(6):338-41. PMID 8046705
- [Background] Buse DC, Reed ML, Fanning KM, Bostic R, Dodick DW, Schwedt TJ, Munjal S, Singh P, Lipton RB. Comorbid and co-occurring conditions in migraine and associated risk of increasing headache pain intensity and headache frequency: results of the migraine in America symptoms and treatment (MAST) study. J Headache Pain. 2020 Mar 2;21(1):23. doi: 10.1186/s10194-020-1084-y. PMID 32122324
- [Background] Headache Classification Committee of the International Headache Society (IHS) The International Classification of Headache Disorders, 3rd edition. Cephalalgia. 2018 Jan;38(1):1-211. doi: 10.1177/0333102417738202. No abstract available. PMID 29368949
- [Background] Edmeads J, Findlay H, Tugwell P, Pryse-Phillips W, Nelson RF, Murray TJ. Impact of migraine and tension-type headache on life-style, consulting behaviour, and medication use: a Canadian population survey. Can J Neurol Sci. 1993 May;20(2):131-7. doi: 10.1017/s0317167100047697. PMID 8334575
- [Background] Kwilasz AJ, Todd LS, Duran-Malle JC, Schrama AEW, Mitten EH, Larson TA, Clements MA, Harris KM, Litwiler ST, Wang X, Van Dam AM, Maier SF, Rice KC, Watkins LR, Barrientos RM. Experimental autoimmune encephalopathy (EAE)-induced hippocampal neuroinflammation and memory deficits are prevented with the non-opioid TLR2/TLR4 antagonist (+)-naltrexone. Behav Brain Res. 2021 Jan 1;396:112896. doi: 10.1016/j.bbr.2020.112896. Epub 2020 Sep 6. PMID 32905811
- [Background] Kato J, Svensson CI. Role of extracellular damage-associated molecular pattern molecules (DAMPs) as mediators of persistent pain. Prog Mol Biol Transl Sci. 2015;131:251-79. doi: 10.1016/bs.pmbts.2014.11.014. Epub 2015 Jan 30. PMID 25744676
- [Background] Parkitny L, Younger J. Reduced Pro-Inflammatory Cytokines after Eight Weeks of Low-Dose Naltrexone for Fibromyalgia. Biomedicines. 2017 Apr 18;5(2):16. doi: 10.3390/biomedicines5020016. PMID 28536359
- [Background] Su M, Ran Y, He Z, Zhang M, Hu G, Tang W, Zhao D, Yu S. Inhibition of toll-like receptor 4 alleviates hyperalgesia induced by acute dural inflammation in experimental migraine. Mol Pain. 2018 Jan-Dec;14:1744806918754612. doi: 10.1177/1744806918754612. Epub 2018 Jan 8. PMID 29310498
- [Background] Gudala K, Bansal D, Vatte R, Ghai B, Schifano F, Boya C. High Prevalence of Neuropathic Pain Component in Patients with Low Back Pain: Evidence from Meta-Analysis. Pain Physician. 2017 Jul;20(5):343-352. PMID 28727698
- [Background] Cant R, Dalgleish AG, Allen RL. Naltrexone Inhibits IL-6 and TNFalpha Production in Human Immune Cell Subsets following Stimulation with Ligands for Intracellular Toll-Like Receptors. Front Immunol. 2017 Jul 11;8:809. doi: 10.3389/fimmu.2017.00809. eCollection 2017. PMID 28744288
- [Background] Graham GG, Scott KF. Mechanism of action of paracetamol. Am J Ther. 2005 Jan-Feb;12(1):46-55. doi: 10.1097/00045391-200501000-00008. PMID 15662292
- [Background] Bjelland I, Dahl AA, Haug TT, Neckelmann D. The validity of the Hospital Anxiety and Depression Scale. An updated literature review. J Psychosom Res. 2002 Feb;52(2):69-77. doi: 10.1016/s0022-3999(01)00296-3. PMID 11832252
- [Background] HAMILTON M. The assessment of anxiety states by rating. Br J Med Psychol. 1959;32(1):50-5. doi: 10.1111/j.2044-8341.1959.tb00467.x. No abstract available. PMID 13638508
- [Background] Bihari B. Bernard Bihari, MD: low-dose naltrexone for normalizing immune system function. Altern Ther Health Med. 2013 Mar-Apr;19(2):56-65. No abstract available. PMID 23594453
- [Background] Younger J, Mackey S. Fibromyalgia symptoms are reduced by low-dose naltrexone: a pilot study. Pain Med. 2009 May-Jun;10(4):663-72. doi: 10.1111/j.1526-4637.2009.00613.x. Epub 2009 Apr 22. PMID 19453963
- [Background] Younger J, Noor N, McCue R, Mackey S. Low-dose naltrexone for the treatment of fibromyalgia: findings of a small, randomized, double-blind, placebo-controlled, counterbalanced, crossover trial assessing daily pain levels. Arthritis Rheum. 2013 Feb;65(2):529-38. doi: 10.1002/art.37734. PMID 23359310
- [Background] Smith JP, Stock H, Bingaman S, Mauger D, Rogosnitzky M, Zagon IS. Low-dose naltrexone therapy improves active Crohn's disease. Am J Gastroenterol. 2007 Apr;102(4):820-8. doi: 10.1111/j.1572-0241.2007.01045.x. Epub 2007 Jan 11. PMID 17222320
- [Background] Cree BA, Kornyeyeva E, Goodin DS. Pilot trial of low-dose naltrexone and quality of life in multiple sclerosis. Ann Neurol. 2010 Aug;68(2):145-50. doi: 10.1002/ana.22006. PMID 20695007
- [Background] Chopra P, Cooper MS. Treatment of Complex Regional Pain Syndrome (CRPS) using low dose naltrexone (LDN). J Neuroimmune Pharmacol. 2013 Jun;8(3):470-6. doi: 10.1007/s11481-013-9451-y. Epub 2013 Apr 2. PMID 23546884
- [Background] Kaufman DW, Kelly JP, Rosenberg L, Anderson TE, Mitchell AA. Recent patterns of medication use in the ambulatory adult population of the United States: the Slone survey. JAMA. 2002 Jan 16;287(3):337-44. doi: 10.1001/jama.287.3.337. PMID 11790213
- [Background] Krenzelok EP, Royal MA. Confusion: acetaminophen dosing changes based on NO evidence in adults. Drugs R D. 2012 Jun 1;12(2):45-8. doi: 10.2165/11633010-000000000-00000. PMID 22530736
- [Background] Prescott LF. Kinetics and metabolism of paracetamol and phenacetin. Br J Clin Pharmacol. 1980 Oct;10 Suppl 2(Suppl 2):291S-298S. doi: 10.1111/j.1365-2125.1980.tb01812.x. PMID 7002186
- [Background] Aurora SK, Papapetropoulos S, Kori SH, Kedar A, Abell TL. Gastric stasis in migraineurs: etiology, characteristics, and clinical and therapeutic implications. Cephalalgia. 2013 Apr;33(6):408-15. doi: 10.1177/0333102412473371. Epub 2013 Mar 5. PMID 23463252
- [Background] Alstadhaug K, Salvesen R, Bekkelund S. 24-hour distribution of migraine attacks. Headache. 2008 Jan;48(1):95-100. doi: 10.1111/j.1526-4610.2007.00779.x. PMID 18184291
- [Background] Pascual J. Clinical benefits of early triptan therapy for migraine. Headache. 2002 Jan;42 Suppl 1:10-7. doi: 10.1046/j.1526-4610.2002.0420s1010.x. PMID 11966859
- [Background] Burch RC, Loder S, Loder E, Smitherman TA. The prevalence and burden of migraine and severe headache in the United States: updated statistics from government health surveillance studies. Headache. 2015 Jan;55(1):21-34. doi: 10.1111/head.12482. Erratum In: Headache. 2015 Feb;55(2):356. PMID 25600719
- [Background] Lipton RB, Scher AI, Kolodner K, Liberman J, Steiner TJ, Stewart WF. Migraine in the United States: epidemiology and patterns of health care use. Neurology. 2002 Mar 26;58(6):885-94. doi: 10.1212/wnl.58.6.885. PMID 11914403
- [Background] Brandes JL. Global trends in migraine care: results from the MAZE survey. CNS Drugs. 2002;16 Suppl 1:13-8. doi: 10.2165/00023210-200216001-00003. PMID 12196035
- [Background] Buse DC, Rupnow MF, Lipton RB. Assessing and managing all aspects of migraine: migraine attacks, migraine-related functional impairment, common comorbidities, and quality of life. Mayo Clin Proc. 2009 May;84(5):422-35. doi: 10.1016/S0025-6196(11)60561-2. PMID 19411439
- [Background] Lipton RB, Hamelsky SW, Dayno JM. What do patients with migraine want from acute migraine treatment? Headache. 2002 Jan;42 Suppl 1:3-9. doi: 10.1046/j.1526-4610.2002.0420s1003.x. PMID 11966858
- [Background] Bigal ME, Serrano D, Buse D, Scher A, Stewart WF, Lipton RB. Acute migraine medications and evolution from episodic to chronic migraine: a longitudinal population-based study. Headache. 2008 Sep;48(8):1157-68. doi: 10.1111/j.1526-4610.2008.01217.x. PMID 18808500